CLINICAL TRIAL: NCT04211402
Title: A Non-Interventional Pilot Study to Explore the Role of Gut Flora in Obsessive-Compulsive Disorder (OCD)
Brief Title: A Non-Interventional Pilot Study to Explore the Role of Gut Flora in Obsessive-Compulsive Disorder
Status: Withdrawn | Type: Observational
Why Stopped: Company shifted focus
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Other Study IDs: PRG-029
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Obsessive-Compulsive Disorder: Patients with obsessive-compulsive disorder
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no intervention for this study

SUMMARY:
This study seeks to correlate microbiome sequencing data with information provided by patients and their medical records.

DETAILED DESCRIPTION:
The goal of this Research Study is to better understand how the genetic information in subject's microbiome correlates to infection with Obsessive-Compulsive Disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, demonstrating that the patient understands the procedures required for the study and the purpose of the study

   a. May be signed by parent or legal guardian in the case of minor or adult unable to provide consent
2. Male or female of all ages
3. OCI greater than or equal to 21

Exclusion Criteria:

1. Refusal to sign informed consent form
2. History of bariatric surgery, total colectomy with ileorectal anastomosis or proctocolectomy.
3. Postoperative stoma, ostomy, or ileoanal pouch
4. Participation in any experimental drug protocol within the past 12 weeks
5. Treatment with total parenteral nutrition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with OCD
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Correlation of Microbiome to Disease via Relative Abundance Found in Microbiome Sequencing | Three years
  Relative abundance of bacterial classes within taxonomic phyla and, more broadly, within their domain will be analyzed by sequencing the gut microbiome. These data will then be categorized with Obsessive-Compulsive Disorder

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Principal Investigator — ProgenaBiome
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD